CLINICAL TRIAL: NCT05672927
Title: Comparison of the Immune Response After Administration of 2 vs. 3 Doses of the FDA-approved 9-Valent HPV Vaccine Among Women 27-45 Years of Age
Brief Title: Comparing Immune Response of 2 vs 3 HPV Doses (27-45 Years Old)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22-0243
Record Dates: First submitted 2022-12-19; First posted 2023-01-05 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Immunization; HPV Infection; Human Papillomavirus
Keywords: HPV vaccination; Gardasil 9; Noninferiority trial
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Vials submitted for assay will be de-identified and labeled only with the study ID number.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Females, 3-dose standard (Active Comparator): Three doses of the 9-valent HPV vaccine to be administered to the comparison group (27-45 years of age) at 0, 2, and 6 months.
  Interventions: Biological: 9-valent HPV vaccine, 3 doses standard timing
- Females, 2-dose alternative (Experimental): Two doses of the 9-valent HPV vaccine to be administered to the experimental group (27-45 years of age) at 0 and 6 months. Additional HPV vaccine dose will be offered after final blood draw at 12 months.
  Interventions: Biological: 9-valent HPV vaccine, 2 doses alternate timing

INTERVENTIONS:
Biological: 9-valent HPV vaccine, 2 doses alternate timing — Evaluate 2 doses of the 9-valent HPV vaccine across a 12-month period following the 1st dose among 27-45-year-old females.
  Arms: Females, 2-dose alternative
Biological: 9-valent HPV vaccine, 3 doses standard timing — This will be the comparison group for the 2-dose group.
  Arms: Females, 3-dose standard

SUMMARY:
The goal of this clinical trial is to compare a 2-dose and 3-dose series of 9vHPV vaccine among 27-45-year-old females to assess if 2 doses elicit a noninferior immune response. Participants will be randomized 1:1 to either the 2-dose group or the 3-dose group and asked to provide 4 blood samples over a period of 12 months. All 2-dose participants will be offered a 3rd dose after the final blood draw,12 months after their initial vaccination.

DETAILED DESCRIPTION:
The investigators are studying an alternate dosing regimen of an approved drug (9vHPV vaccine) in the population for which it is approved. The vaccine is approved for individuals ages 9-45 years old and participants in this study will be 27-45 years of age. The purpose of the study is to examine the immune response of 2 doses of 9vHPV vaccine. The current recommendation is to administer the vaccine in 3 doses (administered at 0, 1-2 months and 6 months) to those 15-45 years of age, but only 2 doses (administered at 0 and 6 months) if the vaccine series is initiated before age 15. The investigators will conduct a randomized study to determine if 2 doses of elicit a similar immune response to that of a standard 3 dose series in individuals 27-45 years of age. Participants in the study group will receive 2 doses of at 0 and 6 months. Participants in the control group will receive 3 doses of 9vHPV vaccine at 0, 2 months, and 6 months. All participants (target accrual n=618) will have 5 mLs of blood drawn at 0, 1, 7, and 12 months. Following the 12-month blood draw, participants randomized to 2-doses will be offered the 3rd dose. Potential participants will be recruited through the University of Texas Medical Branch (UTMB) clinics and surrounding community, and will be screened for inclusion/exclusion criteria. Eligible patients will sign an informed written consent. At their baseline visit, participants will have their blood drawn, be randomized into either the study or control group, and receive their first dose of the HPV vaccine. All participants will receive compensation administered through a ClinCard following each of the 4 blood draws.

ELIGIBILITY:
Inclusion criteria:

1. Females 27-45 years old.
2. Ability to give informed consent.
3. Has not received any prior doses of the HPV vaccine. This will be verified by the person and state registry (Immtrac), as well as the person's electronic medical record.
4. Reliable telephone access for the duration of the project.
5. Can read and speak in either English or Spanish.
6. Identified source of funding for vaccine such as Medicaid, private health insurance, Texas Healthy Women program, etc.
7. Reports consistent use of reliable birth control and plans to continue its use through study month 13.

Exclusion criteria:

1. Currently pregnant or plans to become pregnant or donate eggs in the next 13 months. Any subjects with positive pregnancy tests at the initial visit will be disqualified from the study and advised to seek prenatal care.
2. Has an immunodeficiency or autoimmune disease such as HIV infection, lymphoma, leukemia, lupus, rheumatoid arthritis, inflammatory bowel disease, or other autoimmune condition.
3. Currently receiving treatment or medication that can suppress immune function including radiation therapy, chemotherapy, cyclosporin, leflunomide (Arava), TNF-α antagonists, monoclonal antibody therapies (including rituximab [Rituxan]), intravenous gamma globulin (IVIG), antilymphocyte sera, other therapy known to interfere with the immune response, or systemic corticosteroids (by mouth or intramuscular injection). Those using or have used steroids that are inhaled, placed in the eye, applied on the skin, or injected into the joint/soft tissue will be considered eligible for the study.
4. History of splenectomy
5. Known allergies to any vaccine components, including aluminum, yeast or Benzonase.
6. Febrile at ≥100°F in the 24 hours prior to vaccination. The patients may be rescheduled for a later date.
7. History of thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injections.
8. History of >10 sexual partners in their lifetime at time of enrollment
9. Plans to move out of the Galveston/Houston area in the 13 months following study entry.

Ages: 27 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 618 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Short-term human papillomavirus (HPV) type-specific antibody response for type HPV-6 | Month 1
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-6, measured as number of participants.
Short-term human papillomavirus (HPV) type-specific antibody response for type HPV-6 | Month 7
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-6, measured as number of participants.
Short-term human papillomavirus (HPV) type-specific antibody response for type HPV-6 | Month 12
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-6, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-11 | Month 1
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-11, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-11 | Month 7
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-11, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-11 | Month 12
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-11, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-16 | Month 1
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-16, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-16 | Month 7
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-16, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-16 | Month 12
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-16, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-18 | Month 1
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-18, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-18 | Month 7
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-18, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-18 | Month 12
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-18, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-31 | Month 1
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-31, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-31 | Month 7
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-31, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-31 | Month 12
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-31, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-33 | Month 1
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-33, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-33 | Month 7
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-33, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-33 | Month 12
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-33, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-45 | Month 1
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-45, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-45 | Month 7
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-45, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-45 | Month 12
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-45, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-52 | Month 1
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-52, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-52 | Month 7
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-52, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-52 | Month 12
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-52, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-58 | Month 1
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-58, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-58 | Month 7
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-58, measured as number of participants.
Short-term HPV type-specific antibody response for type HPV-58 | Month 12
  Yes/No for seroconversion, defined as changing from seronegative (antibody titer below established threshold) to seropositive (antibody titer above established threshold) for HPV-58, measured as number of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Abbey B Berenson, MD, PhD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263